

May 15,2023

Attached are the consent documents for the following study: Multi-level effects of a parenting intervention for enhancing Latino youth health behaviors, NCT03517111.

Please find the latest version, dated 04/24/2020, of the following documents in this order:

- Parent Permission (one document for all three arms/conditions)
- Child Assent (one document for all three arms/conditions)
- Parent Consent- Families Preparing the New Generation
- Parent Consent- Realizing the American Dream
- Parent Consent- Families Preparing the New Generation Plus

The FPNG+ Team



#### Dear Parent/Guardian:

We are from the School of Nutrition and Health Promotion and the School of Social Work at Arizona State University. We are studying 6<sup>th</sup>, 7<sup>th</sup>, and 8<sup>th</sup> graders' life experiences such as their diet habits and what happens when they encounter alcohol, tobacco, and other drugs, including personal drug use and their response at times when they get into situations that are risky. In partnership with the **American Dream Academy**, we are inviting families at many schools to help us. If you will be attending a workshop from the American Dream Academy and agreed to participate in our confidential surveys for parents, we are requesting your permission for your child to be part of this research as well.

Three times throughout the project, your child will be asked to fill out a <u>confidential</u> survey. Each survey takes about 45 minutes, and kids will be asked about their diet, what they know about alcohol, tobacco, and other drugs, as well as about personal life experiences with those drugs including whether they have used illegal drugs. All project surveys are <u>voluntary</u>, and youth will <u>not</u> be penalized for deciding not to participate or by withdrawing at any time. Your child will always have a choice to take a survey or not. There is no effect on your child's school work or records. The surveys are <u>confidential</u>. We will only be collecting contact information for tracking and follow-up purposes, or to clarify your diet-related answers if we have questions. Although the contact information form will be part of the survey, once your child has taken the survey and it has been uploaded to the main database, we will save your child's individual information into a separate database from all of the survey answers so that all is left on the survey is just an ID number. So, your child's name will <u>not</u> be included in reports or in any information that goes to teachers or schools. The survey asks questions about diet and attitudes, behaviors, anti-drug norms, and responses to offers of alcohol or drugs and risky behaviors. Your child will receive an incentive such as key chains and Frisbees for each survey completed.

A small number of families will be randomly selected (by chance) to participate in additional optional data collection in their home every time they complete a survey. If you and your child are selected to participate, a study staff member will visit your home at a time when both you and your child are available to measure your child's height, weight, and blood pressure, and to collect a small blood sample from your child's finger (finger prick to get three to four drops of blood) to measure indicators of diabetes and heart disease risk (HbA1c and cholesterol). This visit is optional and voluntary and will take about 90 minutes. Your child will receive \$10 for each visit for a possible total of \$30 (may be paid in cash, physical gift card, or electronic gift card). You do not have to give permission for your child to participate in this additional visit for your child to be part of the larger study. If desired, we will share blood pressure and finger prick results with your child and you during this visit. If we find values that may indicate high blood pressure or elevated risk for diabetes or heart disease, we will give you the values and recommend that you discuss those with your child's doctor. In addition, we will conduct two phone calls where we ask your child about the foods he/she ate the previous day.

By signing below and returning this letter to the school liaison you give your permission for your child to participate in the surveys. Your decision is entirely <u>voluntary</u>. If you choose not to have your child participate, or to withdraw your child at any time, there will be no penalty or negative effect for you or your child. Even if you give your child permission to participate in the program, your child's participation remains voluntary—he or she gets to choose whether or not to take the surveys or to withdraw at any time with no penalty. The results of the study may be published, but your child's name will not be used.

If you have any questions, please call us at 602-496-0700 and we will be happy to answer them. For more information about us, please visit our website at <a href="http://sirc.asu.edu.">http://sirc.asu.edu.</a> If you have any questions regarding your child's rights as a research subject, or if you feel that your child has been placed at risk, please contact the Chair of the Human Subjects Institutional Review Board, through the ASU Research Compliance Office, at (480) 965-6788.

Thank you for your consideration!

Sincerely,

Sonia Vega-López, Ph.D. Principal Investigator, ASU

# Permission for my child

Derent's signature:

- o YES, my child has permission to participate in the surveys.
- o NO, my child does not have permission to participate in the surveys.

By signing below, you are giving your permission for **your child** to participate in the surveys.

Parent's signature:

Date:

Additional data collection at home and by phone- Permission for my child

YES, my child has permission to participate to participate in the collection of additional data in the home and by phone to measure their height, weight, and blood pressure, to collect a finger prick blood

sample, and to complete two phone calls about the foods he/she eats.

o NO, my child does not have permission to participate in the collection of additional data.

By signing below, you are giving your permission for **your child** to participate in the additional data collection at your home and by phone.

| raients signature. | C | ontact Information | |
|---|---|---|---|
| Please print the following: | _ | | |
| Parent Name: | | | |
| Fir | st | Middle | Last |
| Address:Street | | City | Zip |
| 0001 | | o.i.y | <u> </u> |
| Phone: | Cell | Email: | |
| Child in 6 <sup>th</sup> , 7 <sup>th</sup> , or 8 <sup>th</sup> Grade Na | ame:<br>First | Middle | Last |
| Child's Date of Birth: | 1 | | |
| Mont | n Dav | r<br>Year | |

Name of Child's School:



Dear Student:

We are from the School of Nutrition and Health Promotion and the School of Social Work at Arizona State University. We are doing research to better understand 6<sup>th</sup>,7<sup>th</sup>, and 8<sup>th</sup> graders' life experiences such as what they eat and what happens when they are exposed to alcohol, tobacco, and other drugs. Schools all around Phoenix, including your school, are helping us. Families who attend the American Dream Academy program are being invited to help us, too. We hope this research will help us find out ways to help kids like you to stay drug free and eat a healthy diet.

You are being invited to help us by filling out three confidential surveys throughout the year. Each survey takes about 45 minutes, and you will be asked about diet, alcohol, tobacco, and drugs. The surveys are voluntary. Your parent/guardian has given permission for you to fill it out, but you get to decide if you want to take the survey. We will only collect contact information for tracking and follow-up purposes, or to clarify your diet-related answers if we have questions. So even though the contact information form is part of the survey, once you take the survey and it is uploaded to the main database, we will take out your contact information and put it in a separate database from all of the survey answers so that all that will be left on your survey is just an ID number. After this, your information will be confidential. So, your parents will never find out what answers you choose and neither will your teachers or your school. You will receive a small item, such as a Frisbee or a key chain, as our way to thank you for completing each survey.

A small number of families will also be invited to participate in additional data collection in their home and by phone. If your family is selected, you will be invited to also allow us to measure your height, weight, and blood pressure, and give us a small blood sample from your finger (finger prick—3 to 4 drops). The blood test will help us learn more about indicators of diabetes and heart disease risk. These optional activities will take about 90 minutes. You will receive \$10 for each home visit for a possible total of \$30. These will be paid with cash, physical gift card, or electronic gift card. We will also ask you to complete two phone calls where we will ask you about the foods you ate the day before.

By filling out and signing the form below, you agree to take the survey. You can also indicate whether you would like to participate in the additional data collection activities if your family is selected for those. If you choose not to or if you want to stop at any time, there's no penalty—it won't affect your grade or anything. If you would like to take the survey, please fill in the spaces below and return this letter to your facilitator.

If you have any questions, you can always call us at 602-496-0700 and we will be happy to answer them. For more information, please visit our website at <a href="http://sirc.asu.edu">http://sirc.asu.edu</a>. **Thank you!** 

Sincerely,

Sonia Vega-López, Ph.D., Principal Investigator ASU, Phoenix, AZ

# **Project surveys**

the survey because I want to, and I know that I can stop any time. I can skip any questions I don't want to answer, and I know that deciding not to participate is okay. Signature:\_\_\_\_\_\_Date:\_\_\_\_\_ Additional data collection at home and by phone Please check one of the following options below about additional data collection in your home and by phone: ☐ I DO agree to participate in the collection of additional data in my home to measure my height, weight, and blood pressure, to collect a finger prick blood sample, and to complete two phone calls about the foods I eat. I understand that I may choose not to participate at any time. ☐ I DO NOT agree to participate in the collection of additional data. Signature: Date: Please print: Your Name: Middle Month of birth: Day of birth: **Names of your Parents** or Guardians: First Middle Last

I know I have permission to take the surveys and I know what the questions are about. I going to take

Last

First

Middle



#### Dear Parent:

We are from the School of Nutrition and Health Promotion and the School of Social Work at Arizona State University. We are studying 6<sup>th</sup>,7<sup>th</sup>, and 8<sup>th</sup> graders' life experiences such as their diet habits and what happens when they encounter alcohol, tobacco, and other drugs, including personal drug use and their response at times when they get into situations that are risky. Parents who participate in the American Dream Academy workshops throughout the Valley are helping us. We are requesting your participation in workshops called *Families Preparing the New Generation*. During the workshops, you will learn how to reinforce anti-drug norms that are culturally appropriate, how to help strengthen your children, and how to communicate with your child about sensitive topics such as drug use/abuse and other risky behaviors. The program is specifically designed for parents of 6<sup>th</sup>-8<sup>th</sup> graders, but all parents are invited and welcome to attend.

Three times throughout the academic year, you will be asked to fill out confidential surveys to help us. Each survey takes about 60 minutes. You will be asked about your family practices, family communication, and relationship with your child. All project surveys are voluntary, and there is no impact on your student's schoolwork or academic records. We will only be collecting contact information for tracking and follow-up purposes, or to clarify your diet-related answers if we have questions. Although the contact information form will be part of the survey, once you have taken the survey and it has been uploaded to the main database, we will save your contact information into a separate database from all of the survey answers so that all that is left on the survey is just a unique ID number. People who agree to participate in the surveys will have this unique identification code that links them with their children but not to anyone else. That code will be used throughout the study. Because an identification code is used, your name will not be included on any survey or in any reports. You will receive \$10 for the first survey, \$15 for the second survey, and \$20 for the last survey, to thank you for your time (these may be in cash, physical gift card, or electronic gift card). Parents who attend at least 8 ADA sessions will be eligible to participate in a \$25 gift card raffle. There will be two winners in the AM group, and two in the PM group. Please remember that if you choose not to participate in the research study, you can still attend all of the 2 hour longworkshops.

A small number of participants will be randomly selected (by chance) to participate in additional optional data collection in their home every time they complete a survey. If you are selected to participate, a study staff member will visit your home to measure your height, weight, and blood pressure, and to collect a small blood sample from your finger (finger prick to get three or four drops of blood) to measure indicators of diabetes and heart disease risk (HbA1c and cholesterol). The study staff will also ask permission to inventory the foods you keep in your kitchen. This visit is optional and voluntary and will take about 90 minutes. You do not have to agree to this additional visit to be part of the larger study or to participate in the American Dream Academy workshop. If you choose to participate in these three additional visits, you will receive \$20 for each visit (may be paid in cash, physical gift card, or electronic gift card) for a possible total of \$60 for all visits together. If desired, we will share blood pressure and finger prick results with you during this visit. If we find values that may indicate high blood pressure or elevated risk for diabetes or heart disease, we will give you the values and recommend that you discuss those with you doctor. We also ask your permission to complete two phone calls where we will ask you about the foods you ate the previous day.

By filling out the consent form below, you are telling us that you wish to participate in these parent workshop surveys and whether you would agree to participate in the additional data collection in your home. If you choose not to participate, or if you want to stop at any time, there is no penalty—it won't affect you or your child negatively in any way. Your choice will not affect your student's academic records or schoolwork. If you would like to participate, please fill in the spaces below and return the signed form to your facilitator at this meeting.

If you have any questions at any time, please call us at 602-496-0700, and we will be happy to answer them. For more information about us, please visit our website at <a href="http://sirc.asu.edu">http://sirc.asu.edu</a>. If you have any questions regarding your rights as a research participant, or if you feel that you or your family's personal security has been placed at risk, please contact the Chair of the Human Subjects Institutional Review Board, through the ASU Research Compliance Office, at (480) 965-6788.

| Thank you for vo | ır consideration! |
|------------------|-------------------|
|------------------|-------------------|

Sincerely,

Sonia Vega-López, Ph.D., Principal Investigator Downtown Phoenix Campus, ASU, Phoenix, AZ 85004

#### **PLEASE READ THIS:**

# Project surveys

I agree to participate in the three project surveys but understand that I may choose not to participate at any time. I understand that by filling in the spaces below, the information will be used by project staff to keep research project contact information.

| Signature: | Date: |
|---|---|
| Additional data collection at home an | nd by phone |
| Please check one of the following option | ns below regarding additional data collection in your home: |
| weight, and blood pressure, to collect a | ction of additional data in my home to measure my height, finger prick blood sample, to inventory the foods I keep in my s about the foods I eat. I understand that I may choose not to |
| ☐ I DO NOT agree to participate in the | collection of additional data. |
| Signature: | |

| Do you have a child in 6th, 7th, or 8th gra | ide? | Yes 🔲 | No 🗆 | |
|---|---|---|---|---|
| If yes, select your child's grade (circle | e one): 6th | 7th 81 | th | |
| If you have more than one child in the closest to age 13. | se grades, pleas | se think a | about the one who is | |
| 9 | Contact Informa | ation | | |
| Please print the following: | | | | |
| Your Name:First | Middle | | Last | _ |
| Month of birth: Day of birth: | | | | |
| Address:Street | City | | Zip | |
| Phone: Home Cell | E | Email: | | |
| Child in 6 <sup>th</sup> ,7 <sup>th</sup> , or 8 <sup>th</sup> Grade Name: | t | Middle | Last | |
| Child's Date of Birth: / Month | <i>l</i><br>Day Year | | | |
| Name of Child's School: | | | | |



#### Dear Parent:

We are from the School of Nutrition and Health Promotion and the School of Social Work at Arizona State University. We are studying 6<sup>th</sup>, 7<sup>th</sup>, and 8<sup>th</sup> graders' life experiences such as their diet habits and what happens when they encounter alcohol, tobacco, and other drugs, including personal drug use and their response at times when they get into situations that are risky. Parents who participate in the American Dream Academy workshops throughout the Valley are helping us. We are requesting your participation in workshops called *Realizing the American Dream*. During the workshops, you will learn how to work with your child towards becoming successful in school. The program is specifically designed for parents of 6<sup>th</sup>-8<sup>th</sup> graders, but all parents are invited and welcome to attend.

Three times throughout the academic year, you will be asked to fill out confidential surveys to help us. Each survey takes about 60 minutes. You will be asked about your family practices, family communication, and relationship with your child. All project surveys are voluntary, and there is no impact on your student's schoolwork or academic records. We will only be collecting contact information for tracking and follow-up purposes or to clarify your diet-related answers if we have questions. Although the contact information form will be part of the survey, once you have taken the survey and it has been uploaded to the main database, we will save your contact information into a separate database from all of the survey answers so that all that is left on the survey is just a unique ID number. People who agree to participate in the surveys will have this unique identification code that links them with their children but not to anyone else. That code will be used throughout the study. Because an identification code is used, your name will not be included on any survey or in any reports. You will receive \$10 for the first survey, \$15 for the second survey, and \$20 for the last survey, to thank you for your time (these may be in cash, physical gift card, or electronic gift card). Parents who attend at least 8 ADA sessions will be eligible to participate in a \$25 gift card raffle. There will be two winners in the AM group, and two in the PM group. Please remember that if you choose not to participate in the research study, you can still attend all of the 2 hour long workshops.

A small number of participants will be randomly selected (by chance) to participate in additional optional data collection in their home every time they complete a survey. If you are selected to participate, a study staff member will visit your home to measure your height, weight, and blood pressure, and to collect a small blood sample from your finger (finger prick to get three to four drops of blood) to measure indicators of diabetes and heart disease risk (HbA1c and cholesterol). The study staff will also ask permission to inventory the foods you keep in your kitchen. This visit is optional and voluntary and will take about 90 minutes. You do not have to agree to this additional visit to be part of the larger study or to attend the American Dream Academy workshops. If you choose to participate in these three additional visits, you will receive \$20 (may be paid in cash, physical gift card, or electronic gift card) for each visit for a possible total of \$60 for all visits together. If desired, we will share blood pressure and finger prick results with you during this visit. If we find values that may indicate high blood pressure or elevated risk for diabetes or heart disease, we will give you the values and recommend that you discuss those with you doctor. We also ask your permission to complete two phone calls where we will ask you about the foods you ate the previous day.

By filling out the consent form below, you are telling us that you wish to participate in these parent workshop surveys and whether you would agree to participate in the additional data collection in your home. If you choose not to participate, or if you want to stop at any time, there is no penalty —it won't affect you or your child negatively in any way. Your choice will not affect your student's academic records or schoolwork. If you would like to participate, please fill in the spaces below and return the signed form to your facilitator at this meeting.

If you have any questions at any time, please call us at 602-496-0700, and we will be happy to answer them. For more information about us, please visit our website at <a href="http://sirc.asu.edu">http://sirc.asu.edu</a>. If you have any questions regarding your rights as a research participant, or if you feel that you or your family's personal security has been placed at risk, please contact the Chair of the Human Subjects Institutional Review Board, through the ASU Research Compliance Office, at (480) 965-6788.

# Thank you for your consideration!

Sincerely,

Sonia Vega-López, Ph.D., Principal Investigator Downtown Phoenix Campus, ASU, Phoenix, AZ 85004

#### **PLEASE READ THIS:**

## **Project surveys**

Signature:

| • | ect surveys but understand that I may choose not to hat by filling in the spaces below, the information will be project contact information. |
|---|---|
| Signature: | Date: |

# Additional data collection at home and by phone

Please check one of the following options below regarding additional data collection in your home:

| height, weight, and blood pressure, to collect a finger prick blood sample, to inventory the |
|---|
| foods I keep in my kitchen, and to complete two phone calls about the foods I eat. I |
| understand that I may choose not to participate at any time. |

| DO NOT agree to participate in the collection of a | ıdditional data. |
|----------------------------------------------------|------------------|

| Do you have a child in 6th, 7th, or 8th go | rade? | Yes 🗌 | No 🔲 | |
|---|---|---|---|---|
| If yes, select your child's grade (cire | cle one): 6th | 7th 8 | Bth | |
| If you have more than one child in th closest to age 13. | ese grades, ple | ease think | about the one | e who is |
| 9 | Contact Inform | ation_ | | |
| Please print the following: | | | | |
| Your Name:First | Middle | : | L | ast |
| Month of birth: | Day of birth | : | | |
| Address: | <b></b> | | _ | |
| Street | City | | 2 | <sup>2</sup> ip |
| Phone: Home Cell | | Email: | | |
| Child in 6 <sup>th</sup> -8 <sup>th</sup> Grade Name:<br>First | | Middle | | Last |
| | | Middle | | Luot |
| Child's Date of Birth: / Month | Day Year | | | |
| Name of Child's School: | | | | |



#### Dear Parent:

We are from the School of Nutrition and Health Promotion and the School of Social Work at Arizona State University. We are studying 6<sup>th</sup>,7<sup>th</sup>, and 8<sup>th</sup> graders' life experiences such as their diet habits and what happens when they encounter alcohol, tobacco, and other drugs, including personal drug use and their response at times when they get into situations that are risky. Parents who participate in the American Dream Academy workshops throughout the Valley are helping us. We are requesting your participation in workshops called *Families Preparing the New Generation Plus*. During the workshops, you will learn how to reinforce anti-drug norms that are culturally appropriate, how to help strengthen your children, and how to communicate with your child about sensitive topics such as drug use/abuse and other risky behaviors. You will also learn about strategies to improve the quality of your child's diet. The program is specifically designed for parents of 6<sup>th</sup> - 8<sup>th</sup> graders, but all parents are invited and welcome to attend.

Three times throughout the academic year, you will be asked to fill out confidential surveys to help us. Each survey takes about 60 minutes. You will be asked about your family practices, family communication, and relationship with your child. All project surveys are voluntary, and there is no impact on your student's schoolwork or academic records. We will only be collecting contact information for tracking and follow-up purposes, or to clarify your diet-related answers if we have questions. Although the contact information form will be part of the survey, once you have taken the survey and it has been uploaded to the main database, we will save your contact information into a separate database from all of the survey answers so that all that is left on the survey is just a unique ID number. People who agree to participate in the surveys will have this unique identification code that links them with their children but not to anyone else. That code will be used throughout the study. Because an identification code is used, your name will not be included on any survey or in any reports. You will receive \$10 for the first survey, \$15 for the second survey, and \$20 for the last survey, to thank you for your time (these may be in cash, physical gift card, or electronic gift card). Parents who attend at least 8 ADA sessions will be eligible to participate in a \$25 gift card raffle. There will be two winners in the AM group, and two in the PM group. Please remember that if you choose not to participate in the research study, you can still attend all of the 2 hour longworkshops.

A small number of participants will be randomly selected (by chance) to participate in additional optional data collection in their home every time they complete a survey. If you are selected to participate, a study staff member will visit your home to measure your height, weight, and blood pressure, and to collect a small blood sample from your finger (finger prick to get three to four drops of blood) to measure indicators of diabetes and heart disease risk (HbA1c and cholesterol). The study staff will also ask permission to inventory the foods you keep in your kitchen. This visit is optional and voluntary and will take about 90 minutes. You do not have to agree to this additional visit to be part of the larger study or to participate in the American Dream Academy workshop. If you choose to participate in these three additional visits, you will receive \$20 (may be paid in cash, physical gift card, or electronic gift card) for each visit for a possible total of \$60 for all visits together. If desired, we will share blood pressure and finger prick results with you during this visit. If we find values that may indicate high blood pressure or elevated risk for diabetes or heart disease, we will give you the values and recommend that you discuss those with you doctor. We also ask your permission to complete two phone calls where we will ask you about the foods you ate the previous day.

By filling out the consent form below, you are telling us that you wish to participate in these parent workshop surveys and whether you would agree to participate in the additional data collection in your home. If you choose not to participate, or if you want to stop at any time, there is no penalty—it won't affect you or your child negatively in any way. Your choice will not affect your student's academic records or schoolwork. If you would like to participate, please fill in the spaces below and return the signed form to your facilitator at this meeting.

If you have any questions at any time, please call us at 602-496-0700, and we will be happy to answer them. For more information about us, please visit our website at <a href="http://sirc.asu.edu">http://sirc.asu.edu</a>. If you have any questions regarding your rights as a research participant, or if you feel that you or your family's personal security has been placed at risk, please contact the Chair of the Human Subjects Institutional Review Board, through the ASU Research Compliance Office, at (480) 965-6788.

# Thank you for your consideration!

Sincerely,

Sonia Vega-López, Ph.D., Principal Investigator Downtown Phoenix Campus, ASU, Phoenix, AZ 85004

## **PLEASE READ THIS:**

## **Project surveys**

I agree to participate in the three project surveys but understand that I may choose not to participate at any time. I understand that by filling in the spaces below, the information will be used by project staff to keep research project contact information.

| Signature: | Date: |
|---|---|
| Additional data collection at home and b | oy phone |
| Please check one of the following options by phone: | pelow regarding additional data collection in your home and |
| weight, and blood pressure, to collect a fing | on of additional data in my home to measure my height, ger prick blood sample, to inventory the foods I keep in my bout the foods I eat. I understand that I may choose not to |
| ☐ I DO NOT agree to participate in the col | lection of additional data. |
| Signature: | |

| Do you have a child in 6th, 7th, or 8th grade? Yes ☐ No ☐ | | | |
|---|---|---|---|
| If yes, select your child's grade (circle one): 6th 7th 8th | | | |
| If you have more than one child closest to age 13. | in these grades, ple | ease think about the on | e who is |
| | Contact Infor | <u>mation</u> | |
| Please print the following: | | | |
| Your Name: | Mid | dle | Last |
| Month of birth: | Day of bir | th: | _ |
| Address:Street | City | , | Zip |
| Phone: Home | Cell | Email: | |
| Child in 6 <sup>th</sup> -8 <sup>th</sup> Grade Name: | First | Middle | Last |
| Child's Date of Birth: Month | <i>J J</i> Day Yea | ar | |
| Name of Child's School: | | | |